CLINICAL TRIAL: NCT03892005
Title: A Multi-Centre Post Market Clinical Follow-Up Study of MOTIVATION HIP Total Hip System in Total Hip Arthroplasty
Brief Title: PMCF Study of MOTIVATION HIP System in THA
Status: Suspended | Type: Observational
Why Stopped: No plan to extend CE Mark
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: CSA2018-04H
Record Dates: First submitted 2019-03-08; First posted 2019-03-27 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Total Hip Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MOTIVATION HIP Total Hip System: All study subjects have undergone routine preoperative clinical evaluations prior to their THA, and implanted MOTIVATION HIPTM Total Hip System in accordance to indications and intended use, and appropriate surgical technique(s) will be invited to participate in the study at their first year of postoperative follow up visit, and sign ICF.
  Interventions: Procedure: Total Hip Arthroplasty using MOTIVATION HIP Total Hip System

INTERVENTIONS:
Procedure: Total Hip Arthroplasty using MOTIVATION HIP Total Hip System — To systemically document the clinical safety and performance of the commercially available MOTIVATION HIP Total Hip System in primary THA.

SUMMARY:
This is a retrospective and prospective, multi-center, post-market clinical follow-up study involving orthopedic surgeons skilled in THA and experienced implanting the study device system.

DETAILED DESCRIPTION:
The objective of this study is to obtain implant survivorship and clinical outcomes data for the commercially available MOTIVATION HIP Total Hip System used in primary total hip arthroplasty (THA).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years old, inclusive.
* Had a primary unilateral or bilateral (simultaneous or staged) THA based on physical exam and medical history, including diagnosis of severe hip pain and disability.
* Had received MOTIVATION HIPTM Total Hip System per the approved indications for use for the THA.
* No history of previous prosthetic replacement device of any type, including surface replacement arthroplasty, endoprosthesis, etc. of the affected hip joint(s) beside investigational product.
* Willing and able to provide written informed consent by signing and dating the EC approved informed consent form.
* Willing and able to complete scheduled follow-up evaluations..

Exclusion Criteria:

* The patient is:

  * A prisoner
  * Mentally incompetent or unable to understand what participation in the study entails
  * A known alcohol or drug abuser
  * Anticipated to be non-compliant

    * Has a neuromuscular disorder, vascular disorder or other conditions that could contribute to prosthesis instability, prosthesis fixation failure or complications in postoperative care.
    * Has a neurologic condition in the ipsilateral or contralateral limb which affects lower limb function.
    * Has a diagnosed systemic disease that could affect his/her safety or the study outcome.
    * Known to be pregnant.
    * Has an active or latent infection in or about the affected hip joint or an infection distant from the hip joint that may spread to the hip hematogenously.
    * Insufficient bone stock to fix the component. Insufficient bone stock exists in the presence of metabolic bone disease (i.e., osteoporosis), cancer, and radiation.
    * Osteoradionecrosis in the affected hip joint.
    * Known sensitivity or allergic reaction to one or more of the implanted materials.
    * Known local bone tumors and/or cysts in the operative hip.
    * Body Mass Index (BMI) > 40.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population are patients who have received MOTIVATION HIPTM Total Hip System for their primary THA and meet the Patient Selection Criteria outlined in the protocol.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Implant survivorship based on revision rate | 10 years
  Implant survivorship will be assessed using a Kaplan-Meier analysis. Data will be considered right-censored for all subjects that do not have a device related failed. For subjects who are lost-to-follow up, their last available clinical visit will be considered as the censored date. For subjects who died during the study, their death date will be used as the censored date. The survivorship point estimate and 95% confidence interval about the point estimate will be calculated for each follow up visit (1 year, 2 years, 3 years, 5 years, 7 years and 10 years).

SECONDARY OUTCOMES:
Functional outcome based on Harris Hip Score | 10 years
  Harris Hip Score is a clinician-based outcome measure consisting of 4 subscales. The first is pain, which measures pain severity (44 points); function, which is made up of daily activities and gait (47 points); the absence of deformity, which is a subscale that measures hip flexion, adduction, internal rotation, leg length discrepancy and range of motion measures.(4 points), and range of motion (5 points). The scores range from 0-100 with higher scores representing less dysfunction and better outcomes.
Quality of life based on EQ-5D questionnaire | 10 years
  EQ-5D is a standardized measure of health-related quality of life states consisting of 5 dimensions, namely mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The EQ-5D-5L version was used in the study. Each dimension has 5 responses recording 5 levels of severity (no problems/slight problems/moderate problems/severe problems or extreme problems). The responses to the EQ-5D dimensions are used to obtain a single EQ-5D index value where 1 represents full health and 0 represents death. The questionnaire also includes a vertical, visual analogue scale (EQ VAS) for the respondents to record their self-rated health where the 2 extreme ends of the scale are labelled as 'Best imaginable health state' and 'Worst imaginable health state' respectively.
Safety assessment | 10 years
  Summarize the category, incidence and frequency of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Yuchang Zhu, Professor, Principal Investigator — Shanghai Tenth Hospital
Locations (1):
- Shanghai Tenth Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No